CLINICAL TRIAL: NCT00178256
Title: A Phase I/II Clinical Trial Of Pulsed Paclitaxel And Daily Thoracic Radiotherapy For Inoperable (Stage I/II) Or Unresectable (Stage III) Lung Cancers
Brief Title: Pulsed Paclitaxel And Daily Thoracic Radiotherapy For Inoperable (Stage I/II) Or Unresectable Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Yuhchyau Chen, Principal Investigator, University of Rochester
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URCC 1597
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2014-01-30 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Radiotherapy

ARMS (4):
- 1st dose cohort 15mg/m2 taxol plus RT (Experimental): 15 mg/m2 Paclitaxel On Mondays, Wednesdays, and Fridays, paclitaxel infusion will begin early in the morning and complete before 10:30 am.
  On Monday, Tuesday, Wednesday, Thursday, Friday Thoracic XRT will be given in late afternoon, after 4:00 PM, if possible
  Interventions: Drug: Paclitaxel; Procedure: Radiation Therapy
- 2nd dose cohort20 mg/m2 taxol plus daily RT (Experimental)
  Interventions: Drug: Paclitaxel; Procedure: Radiation Therapy
- 3rd Dose Cohort --25mg/m2 taxol plus RT (Experimental)
  Interventions: Drug: Paclitaxel; Procedure: Radiation Therapy
- Phase II Arm --20mg/m2 taxol plus RT (Experimental)
  Interventions: Drug: Paclitaxel; Procedure: Radiation Therapy

INTERVENTIONS:
Drug: Paclitaxel — On Mondays, Wednesdays, and Fridays, paclitaxel infusion will begin early in the morning and complete before 10:30 am.
Procedure: Radiation Therapy — Thoracic XRT will be given in late afternoon, after 4:00 PM, if possible

SUMMARY:
A treatment study is being conducted by the University of Rochester Cancer Center (URCC) in which patients with non-small cell lung cancer will be treated with radiation therapy and a drug called paclitaxel. Paclitaxel is a natural product with anticancer properties. The first purpose of this study is to determine the dose of paclitaxel which, when given in combination with radiation therapy, will provide the greatest effect have the least side effects. To determine this, patients will be put on the study in groups of 3. The dose for each additional group will be higher than the previous dose until the maximum tolerated dose is reached. The second purpose is to determine if radiation therapy with paclitaxel is more effective in treating lung cancer than radiation therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed lung cancer, excluding small cell carcinoma
* Inoperable stage I (T1-2N0) and II (T1-2N1, T3N0) disease, or stage IIIA (T3N1 andT1-3N2M0) and IIIB (TxN3M0, T4NxM0) diseases according to the American Joint Committee of Cancer criteria 1998
* The primary tumor must be radiographically measurable.
* Age > 18.
* Karnofsky performance status > 70.
* FEV1 sufficient for patients to tolerate radiation therapy which is at the discretion of the radiation oncologist, usually > 800 ml
* Labs: WBC > 3000; platelet count > 100,000; serum creatinine < 1.5 mg/dl or creatinine clearance >60 ml/min.
* Laboratory values must be obtained < 3 weeks prior to registration.
* A signed informed consent.
* Patients who failed prior chemotherapy are eligible. Patients with prior radiotherapy to the chest region are eligible as long as the normal tissue tolerance is not violated by repeat radiotherapy.

Exclusion Criteria:

* Patients with medical contraindication to chemotherapy or radiotherapy.
* Patients with myocardial infarction within the preceding six months or symptomatic heart disease, including uncontrolled or unstable angina, uncontrolled congestive heart failure, and uncontrolled arrhythmia.
* Women who are pregnant.
* Patients with small cell carcinoma or mesothelioma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 1998-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuhchyau Chen, MD, Ph.D, Principal Investigator — Universtiy of Rochester, Dept of Radiation Oncology
Locations (1):
- University of Rochester, Dept. Radiation Oncology, Rochester, New York, United States

REFERENCES:
- [Result] Chen Y, Pandya K, Keng PC, Johnstone D, Li J, Lee YJ, Smudzin T, Okunieff P. Phase I/II clinical study of pulsed paclitaxel radiosensitization for thoracic malignancy: a therapeutic approach on the basis of preclinical research of human cancer cell lines. Clin Cancer Res. 2003 Mar;9(3):969-75. PMID 12631594

RESULTS

PARTICIPANT FLOW:
Groups:
- First Dose Cohort (15mg/m2 Taxol) MWF and Daily RT; Second Dose Cohort (20mg/m2 Taxol) MWF and Daily RT: On Mondays, Wednesdays, and Fridays, paclitaxel infusion will given. On Monday, Tuesday, Wednesday, Thursday, Friday Thoracic XRT will be given.
  A minimum of three patients will be assigned at each dose level.
  If no DLTs are observed then the next three patients enrolled will receive a dose of 5 mg/m2 per dose more than the previous group.
  If one or two instances of DLT are observed then an additional three patients will be tested at the same dose. If DLT is observed in at most two of six patients then dose escalation will continue in the next three patients enrolled.
  Dose-limiting toxicity (DLT) is defined as grade 4 hematologic toxicity, or grade 3 and 4 non-hematologic toxicity excluding nausea and vomiting according to RTOG and Cooperative Group common toxicity criteria. The adverse event must be related to the treatment (paclitaxel or radiation) to be considered a DLT
- Third Dose Cohort (25mg/m2 Taxol) MWF and Daily RT: A minimum of three patients will be assigned at each dose level.
  If no DLTs are observed then the next three patients enrolled will receive a dose of 5 mg/m2 per dose more than the previous group.
  If one or two instances of DLT are observed then an additional three patients will be tested at the same dose. If DLT is observed in at most two of six patients then dose escalation will continue in the next three patients enrolled.
  Dose-limiting toxicity (DLT) is defined as grade 4 hematologic toxicity, or grade 3 and 4 non-hematologic toxicity excluding nausea and vomiting according to RTOG and Cooperative Group common toxicity criteria. The adverse event must be related to the treatment (paclitaxel or radiation) to be considered a DLT
- Phase II Group (20mg/m2 Taxol): Once the MTD has been determined and confirmed with a total of six patients, up to 19 additional patients with measurable disease will be enrolled at that dose in order to obtain estimates of response rate and more information about toxicity Phase II enrollment will be in two stages. Initially 9 or 12 patients (depending on how many were tested at the MTD dose in the Phase I study) will be tested, for a total of 15 patients at the MTD. If fewer than 4 responses are observed, the study will end with 90% confidence that the true response rate is no greater than 40%, which is the minimum clinically interesting response rate.
  If four or more responses are observed, additional patients will be enrolled to obtain 25 evaluable patients at the MTD. This will allow estimation of the true response rate and toxicity rates with standard errors of no more than 0.1.
Period: Overall Study
Arm/Group | First Dose Cohort (15mg/m2 Taxol) MWF and Daily RT | Second Dose Cohort (20mg/m2 Taxol) MWF and Daily RT | Third Dose Cohort (25mg/m2 Taxol) MWF and Daily RT | Phase II Group (20mg/m2 Taxol)
Started | 10 | 7 | 6 | 18
Completed | 6 | 6 | 6 | 16
Not Completed | 4 | 1 | 0 | 2
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 1
Not completed — Cancer progression | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Daily RT Plus Chemo on MWF: Paclitaxel On Mondays, Wednesdays, and Fridays, paclitaxel infusion will begin early in the morning and complete before 10:30 am.
  On Monday, Tuesday, Wednesday, Thursday, Friday Thoracic XRT will be given in late afternoon, after 4:00 PM, if possible
  Radiation Therapy : Thoracic XRT will be given in late afternoon, after 4:00 PM, if possible
  Paclitaxel : On Mondays, Wednesdays, and Fridays, paclitaxel infusion will begin early in the morning and complete before 10:30 am.
Arm/Group | Daily RT Plus Chemo on MWF
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Define the Maximum Tolerated Dose (MTD) Using This Dose Schedule.
Time Frame: 5 years
Measure: Number; unit: Percentage subj w dose limiting toxicity
Groups:
- 1st Dose Cohort 15mg/m2 Taxol Plus RT: 15 mg/m2 Paclitaxel On Mondays, Wednesdays, and Fridays, paclitaxel infusion will begin early in the morning and complete before 10:30 am.
  On Monday, Tuesday, Wednesday, Thursday, Friday Thoracic XRT will be given in late afternoon, after 4:00 PM, if possible
  Paclitaxel: On Mondays, Wednesdays, and Fridays, paclitaxel infusion will begin early in the morning and complete before 10:30 am.
  Radiation Therapy: Thoracic XRT will be given in late afternoon, after 4:00 PM, if possible
Arm/Group | 1st Dose Cohort 15mg/m2 Taxol Plus RT | 2nd Dose cohort20 mg/m2 Taxol Plus Daily RT | 3rd Dose Cohort --25mg/m2 Taxol Plus RT
Number analyzed (Participants) | 10 | 7 | 6
Percentage subj w dose limiting toxicity | 20 | 28.6 | 33.3

2. Secondary Outcome: Median Survival
Description: This is median survival for all subjects enrolled.
Time Frame: 86 months
Measure: Median (Full Range); unit: months
Groups:
- All Pts Enrolled Daily RT Plus Chemo on MWF: Paclitaxel On Mondays, Wednesdays, and Fridays, paclitaxel infusion will begin early in the morning and complete before 10:30 am.
  On Monday, Tuesday, Wednesday, Thursday, Friday Thoracic XRT will be given in late afternoon, after 4:00 PM, if possible
  Radiation Therapy : Thoracic XRT will be given in late afternoon, after 4:00 PM, if possible
  Paclitaxel : On Mondays, Wednesdays, and Fridays, paclitaxel infusion will begin early in the morning and complete before 10:30 am.
Arm/Group | All Pts Enrolled Daily RT Plus Chemo on MWF
Number analyzed (Participants) | 41
months | 10.2 [1.4 to 85.6]

ADVERSE EVENTS:
Arm/Group | All Subjects Enrolled
Serious Adverse Events (participants affected / at risk) | 7/41
Other Adverse Events (participants affected / at risk) | 3/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects Enrolled (N=41)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Adult Respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infection (Infections and infestations) | 1 (1) — community acquired pneumonia
Thromboembolic event (Vascular disorders) | 1 (1) — pulmonary embolism
bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Pathology showed this to be unrelated to the chemotherapy
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects Enrolled (N=18)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Esophagitis (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes